CLINICAL TRIAL: NCT03728036
Title: A Temporal Analysis of the Robustness of Hemiplegic Gait and Standing Balance Early After sTroke - the TARGET Research Project
Brief Title: What do Stroke Survivors Actually Learn When Regaining Walking Ability After Stroke? The TARGET Phase I Study
Acronym: TARGET
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Jonas Schröder, Principle investigator, PhD researcher, Universiteit Antwerpen
Other Study IDs: JS-1; 1S64819N (Other Grant/Funding Number: Fonds Wetenschappelijk Onderzoek (Brussel, Flanders))
Record Dates: First submitted 2018-10-24; First posted 2018-11-01 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Stroke; Paresis; Gait, Hemiplegic
Keywords: walking; recovery; compensation
MeSH Terms: conditions — Stroke; Paresis; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: conventional rehabilitation — The investigated cohort will be exposed to 'standard care' including conventional rehabilitation therapy.

SUMMARY:
Phase I: Exploring what stroke survivors exactly learn when recovering the ability to stand and walk.

DETAILED DESCRIPTION:
GENERAL:

Pre-clinical research has pointed towards a time window of enhanced responsiveness to therapy early after stroke. For example, training has led to substantial recovery if initiated 5 or 14, but not 30 days post-stroke in a rodent model (Biernaski 2004). It is suggested that this early period is characterized by heightened levels of plasticity and that training can exploit this leading to improved outcome. The typically observed non-linear recovery pattern in stroke survivors (Kwakkel 2004) might suggest that similar mechanisms are induced in the human brain, however clinical research on this is disappointingly sparse.

In two closely inter-related phases, we aim to examine the biomechanical changes related to walking recovery in general (Phase I) and the specific effects of robot-assisted training (Phase II). By that, we aim to detect a time window in stroke survivors which resembles the same characteristics as observed in animal models. To initiate gait training at an early stage, when patients usually present severe weakness and balance deficits, a mobile exoskeleton is used which is developed to provide intensive walking practice.

OBJECTIVES:

(I.a) Is there a distinct time window of behavioral restitution (i.e., returning towards pre-stroke movement patterns) underlying early walking recovery?

(I.b) Are improvements in standing and walking throughout the first 6 months post-stroke explained by behavioral restitution or learning to use compensation strategies?

ELIGIBILITY:
Inclusion Criteria:

* First-ever, MRI- or CT-confirmed, ischemic or hemorrhagic, anterior circulation stroke
* Age: 18 - 90 years
* Baseline assessments within the first 14 days after stroke onset
* Weakness of the lower limb (NIHSS item >0 at 72 hours post-stroke)
* Pre-morbid independence in activities of daily living (mRS </=2) and gait (FAC >3)
* Able to communicate and comprehend
* Sufficient motivation to participate
* Provided a written informed consent

Exclusion Criteria:

* No other neurological condition affecting motor functions of the lower limbs
* Pre-existing musculoskeletal impairment severely affecting the gait pattern

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the neurology department of the Antwerp University Hospital after acute stroke will be contacted and asked to participate. Information about the study's aim will be provided with a clear understanding of what is expected from the participant. If the patient express willingness to enter the study, the examination on in- and exclusion criteria will be performed. If the patient is considered eligible, an informed consent will be signed.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Categories | 12 weeks post-stroke]
  This scale indicates the ability to walk independently and serves as the primary outcome measure.

SECONDARY OUTCOMES:
Trunk Control Test - item sitting balance | Baseline (0-1 week post-stroke)
  Sitting balance is part of the prognostic model used to stratify patients at baseline.
  Scoring: 0 - 1 (able to sit independently without support of the legs or trunk 30 seconds)
Motricity Index - subscale lower limb | Baseline (0-1 week post-stroke), 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  Strength of major muscle groups of the paretic lower limb is assessed. At baseline this is part of the prognostic model used to stratify patients.
  Scoring: This scale is scored from 0 (no muscle activity) to 99 (normal strength over full range of motion in hip flexors, knee extensors and ankle dorsiflexors).
Fugl Meyer Motor Assessment - subscale lower limb | Baseline (0-1 week post-stroke), 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  This scale measures the level of of selective control of muscles of the paretic lower limb.
  Scoring: This scale is scored from 0 (no reflex activity) to 34 (volitional movement out of synergism).
Berg Balance Scale - item standing unsupported | Baseline (0-1 week post-stroke), 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  This item of the BBS indicates the ability to stand independently and therefore reflects the process of functional walking recovery within the first 6 months post-stroke.
  Scoring: This scale includes 5 levels (0-4), ranging from "unable to stand 30 seconds unassisted" (0) to "able to stand safely 2 minutes" (5).
Functional Ambulation Categories | Baseline (0-1 week post-stroke), 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  This scale indicates the ability to walk independently and therefore reflects the process of functional walking recovery within the first 6 months post-stroke.
  Scoring: This scale includes 6 levels (0-5), ranging from "nonfunctional ambulation" (0) to "ambulate independently, on level and non-level surfaces including stairs and inclines" (5).
Kinetic analyses of standing balance & gait | 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  Dual-force plate measurements are able to indicate the adopted control strategies for standing balance and walking. These analyses are used to distinguish between behavioral restitution and the use of compensation strategies.
EMG analyses of standing balance & gait | 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  EMG analyses will be performed to gain insights in the muscle recruitment of patients during standing and walking. These analyses are used to distinguish between behavioral restitution and the use of compensation strategies.
Spatio-temporal analyses of gait | 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke.
  Assessing comfortable (self-selected) speed and spatial/temporal symmetry of gait over a short distance.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Schröder, PhD Student, Principal Investigator — Dept. Rehabilitation Sciences & Physiotherapy, University of Antwerp, Belgium; Wim Saeys, Prof. Dr., Study Director — Dept. Rehabilitation Sciences & Physiotherapy, University of Antwerp, Belgium; Steven Truijen, Prof. Dr., Study Chair — Dept. Rehabilitation Sciences & Physiotherapy, University of Antwerp, Belgium; Gert Kwakkel, Prof. Dr., Study Chair — Dept. Rehabilitation Medicine, VU University Medical Center, Amsterdam, Netherlands
Locations (3):
- Belgium (3):
  - Antwerp University Hospital, Antwerp
  - RevArte Rehabilitation Hospital, Antwerp
  - GZA Ziekenhuis - campus St Augustinus & Campus St Vincentius, Wilrijk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroder J, Saeys W, Embrechts E, Hallemans A, Yperzeele L, Truijen S, Kwakkel G. Recovery of Quiet Standing Balance and Lower Limb Motor Impairment Early Poststroke: How Are They Related? Neurorehabil Neural Repair. 2023 Aug;37(8):530-544. doi: 10.1177/15459683231186983. Epub 2023 Aug 19. PMID 37596887